CLINICAL TRIAL: NCT02475447
Title: A Phase 2 Multicenter Study to Evaluate the Safety, Pharmacokinetics and Preliminary Efficacy of Asimadoline in Adult Subjects With Pruritus Associated With Atopic Dermatitis
Brief Title: Safety, Pharmacokinetics and Preliminary Efficacy of Asimadoline in Pruritus Associated With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tioga Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ASMP2006
Record Dates: First submitted 2015-02-10; First posted 2015-06-18 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Pruritus; Atopic Dermatitis
MeSH Terms: conditions — Pruritus; Dermatitis, Atopic | interventions — asimadoline; Clinical Coding

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo-matched tablets twice daily for 4 weeks.
  Interventions: Drug: Placebo
- Asimadoline (Experimental): Asimadoline tablets twice daily (5 mg total daily dose) for 8 weeks.
  Interventions: Drug: Asimadoline

INTERVENTIONS:
Drug: Asimadoline — kappa-opioid receptor agonist
  Other Names: No brand name, serial number and code name
  Arms: Asimadoline
Drug: Placebo — placebo-matched control
  Other Names: No brand name, serial number and code name
  Arms: Placebo

SUMMARY:
Kappa-opioid receptors mediate the sensation of itch in animals and humans. Asimadoline is an orally active, selective kappa-opioid receptor agonist and has demonstrated efficacy in several preclinical pruritus models. The purpose of this Phase 2 study is to evaluate the safety, tolerability and clinical efficacy of asimadoline in patients with pruritus associated with atopic dermatitis.

DETAILED DESCRIPTION:
Asimadoline has been administered to over 1900 human subjects or patients in clinical trials and exhibits an acceptable safety profile. Due to its high selectivity for the kappa-opioid receptor, asimadoline does not produce mu-opioid like side-effects. Results from preclinical models indicate asimadoline significantly reduces the frequency of scratching induced by pruritic agents. This double-blind placebo-controlled clinical study is designed to evaluate the safety, tolerability and clinical efficacy of asimadoline in patients with pruritus associated with atopic dermatitis.

ELIGIBILITY:
Main Inclusion Criteria:

1. Signed informed consent and must be able and willing to follow study procedures and instructions
2. Male or female subject aged 18 years or older (no upper age limit)
3. Established clinical diagnosis of atopic dermatitis for at least 6 months
4. Itching Visual Analog Scale (VAS) average worst itching score of at least 40 mm on a 100 mm scale
5. Female subject of childbearing potential and male subject of procreative capacity agree to use an effective method of contraception for the duration of the study

Main Exclusion Criteria:

1. Pregnant, attempting to conceive, or nursing
2. Received phototherapy (ultraviolet B, psoralen plus ultraviolet A) within the previous 4 weeks
3. Received treatment with any of the following within the previous 2 weeks:

   - Topical or oral immunosuppressants or calcineurin inhibitors, sedating anti-histamines or anti-histamines taken for pruritus treatment, prescription topical corticosteroid creams or ointments, any other oral or topical steroids, aprepitant, naltrexone, pregabalin, gabapentin, or tricyclic antidepressants, or any other medications that, in the investigator's judgement, could affect the subject's pruritus or atopic dermatitis, and that are not specified below

   OR taking any of the following and has not been on stable use for at least the previous 4 weeks:

   - Non-prescription topical hydrocortisone creams or ointments, lotions, moisturizers, emollients, bath oil treatments, non-sedating oral anti-histamines being taken for allergy treatment, selective serotonin reuptake inhibitor (SSRI) antidepressants.
4. Currently participating in other investigational clinical studies or having received investigational drugs in a clinical research study within the previous 3 months. Subjects currently enrolled in an observational study are eligible for participation in this study, however subjects must not enroll in a new observational study during the course of their participation in this study
5. Pruritus due to conditions other than atopic dermatitis (e.g., hepatitis, biliary cirrhosis, scabies) or due to medications known to cause pruritus
6. Acute illnesses, uncontrolled or unmanaged diabetes or thyroid disease, decompensated heart failure, cirrhosis or liver failure, chronic kidney disease, or uncontrolled psychiatric disease
7. Evidence or treatment of malignancy (other than localized basal cell cancer, squamous cell skin cancer, or cancer in situ that has been resected) within the previous 5 years
8. History of HIV infection
9. History of alcohol or drug abuse within the past 3 years
10. Diseases or conditions that could, in the opinion of the investigator, interfere with the assessment of safety and efficacy of the study drug and compliance of the subject with study visits/procedures (e.g. exacerbation of multiple sclerosis or other comorbid conditions)
11. Use of any product that acts as an inhibitor of P-glycoprotein (P-gp) or as a P-gp substrate (with the exception of topical ketoconazole product for skin or scalp) within the previous 4 weeks
12. Known allergy to asimadoline or its drug components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Participants will be followed for the duration of the study, an expected 12 weeks

SECONDARY OUTCOMES:
Change from Baseline in Worst Itching Severity using a Visual Analog Scale | 4 weeks
Maximum observed plasma drug concentration (Cmax) | 0.5, 0.75, 1, 1.5, 2, 3, 5, 6 and 8 hours after dosing
Time to reach Cmax in plasma (Tmax) | 0.5, 0.75, 1, 1.5, 2, 3, 5, 6 and 8 hours after dosing
Area under the plasma concentration-versus-time curve (AUC) from the time of the dose to the end of the 12-hour dosing interval | 0.5, 0.75, 1, 1.5, 2, 3, 5, 6 and 8 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Dawn McGuire, MD FAAN, Study Director — Tioga Pharmaceuticals, Inc.
Locations (22):
- United States (22):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Axis Clinical Research, Los Angeles, California
  - Tory Sullivan, MD PA, North Miami Beach, Florida
  - Park Avenue Dermatology, Orange Park, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Northwest Clinical Trials, Boise, Idaho
  - Sneeze, Wheeze and Itch Associates, LLC, Normal, Illinois
  - Forefront Dermatology, Carmel, Indiana
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - The Dermatology Group, Verona, New Jersey
  - Corning Center for Clinical Research, Corning, New York
  - UNC Dermatology and Skin Cancer Center, Chapel Hill, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Department of Dermatology, Philadelphia, Pennsylvania
  - Temple Itch Center, Philadelphia, Pennsylvania
  - Radiant Research, Inc., Anderson, South Carolina
  - Medical Research South, Charleston, South Carolina
  - National Allergy and Asthma Research, LLC, North Charleston, South Carolina
  - Dermatology Treatment and Research Center, PA, Dallas, Texas
  - Sylvana Research Associates, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No